CLINICAL TRIAL: NCT06415708
Title: Obinutuzumab Combined With Bendamustine in the Treatment of Mature B-cell Lymphoma: an Open-label, Multicenter Study
Brief Title: Obinutuzumab Combined With Bendamustine in the Treatment of Mature B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDHBcell2023
Record Dates: First submitted 2024-03-04; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-01

CONDITIONS: B Cell Lymphoma
Keywords: Obinutuzumab; Bendamustine
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab Combined With Bendamustine (Experimental)
  Interventions: Drug: Obinutuzumab Combined With Bendamustine

INTERVENTIONS:
Drug: Obinutuzumab Combined With Bendamustine — The treatment is divided into two phases: induction therapy and maintenance therapy Induction therapy: 6 cycles of obinutuzumab (1000 mg, IV) on Days 1, 8, and 15 of Cycle 1 and on Day 1 of Cycles 2-6 (28 days/cycle). Bendamustine (90 mg/m2, IV) on Days 1 and 2 of Cycles 1-6.
  Maintenance therapy: Patients who achieved at least a partial response after 6 months of induction therapy were eligible to enter the maintenance phase, during which obinutuzumab (1000 mg, IV) was administered every 2 months for 2 years.

SUMMARY:
This is a prospective, single-center, single-arm clinical study to evaluate the efficacy and safety of maintenance therapy with obinutuzumab for 2 years in patients ≥ 18 years of age with newly diagnosed mature B-cell lymphoma (including follicular lymphoma[FL], marginal zone cell lymphoma[MZL] , waldenström macroglobulinemia[WM], hairy-cell leukemia variant[HCL-v]) who achieved ≥ PR after 6 cycles of obinutuzumab in combination with bendamustine.

DETAILED DESCRIPTION:
This study will explore whether induction therapy with obinutuzumab in combination with bendamustine followed by maintenance therapy with obinutuzumab in treatment-naïve patients with mature B-cell lymphoma will improve the prognosis of patients with this type of indolent mature B-cell lymphoma and the efficacy and safety of this regimen in different lymphoma subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, sign informed consent and comply with the study trial protocol
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
4. FL (grade 1 - 3a), MZL, WM, HCL-v with histological documentation of CD20 positivity
5. Systemic therapy as assessed by the investigator based on tumor size and/or GELF criteria
6. Histological confirmation of MZL. For splenic marginal zone lymphoma (SMZL) for which splenic histological specimens cannot be obtained, it is required to meet the minimum diagnostic criteria for SMZL and rule out any other type of small B-cell lymphoma, that is, it is required to confirm the diagnosis of MZL. If the patient had gastric extranodal MZL with symptoms: H. pylori-negative primary lesion or re-lesion after local therapy (i.e., surgery or radiation therapy), the investigator judged whether treatment was required, and if H. pylori-positive, stable disease, progression, or recurrence after antibiotic treatment, the investigator judged whether treatment was required
7. Waldenström macroglobulinemia,lymphoplasmacytic lymphoma,WM/LPL(WM/LPL): meets the diagnostic criteria for WM/LPL and is indicated for treatment (meets at least one of the following conditions): symptomatic hyperviscosity; symptomatic peripheral neuropathy; amyloidosis; cold agglutinin disease; cryoglobulinemia; disease-related cytopenias (Hb < 100 g/L, PLT < 100 × 109/L); giant lymph nodes; those with systemic symptoms: persistent for two weeks/recurrent fever (above 38℃) and not caused by infection, or night sweats and/or weight loss > 10% within 6 months; rapid disease progression, such as lymph node enlargement of more than 50% within 2 months, and/or absolute doubling time of peripheral blood lymphocytes < 6 months, and/or rapid decrease in hemoglobin or platelets due to non-autoimmune causes
8. HCL-v: Meet the WHO diagnostic criteria (4th Edition, 2016), and treatment is indicated
9. At least one two-dimensional measurable lymph node lesion (maximum diameter > 1.5 cm by CT scan or MRI), or at least one two-dimensional measurable extranodal lesion (maximum diameter > 1.0 cm by CT scan or MRI)
10. Life expectancy ≥ 3 months
11. Adequate blood function (except for abnormalities considered by the investigator to be due to the underlying disease of lymphoma), defined as follows: hemoglobin ≥ 7 g/dL absolute neutrophil count ≥ 1.0 × 10^9/L platelet count ≥ 50 × 10^9/L
12. Normal laboratory values: creatinine clearance ≥ 30 mL/min AST or ALT ≤ 2.5 x upper limit of normal (ULN) Serum bilirubin ≤ 2 x ULN (≤ 3 x ULN for patients with Gilbert's syndrome) measured or estimated according to institutional standard methods
13. For men who are not surgically sterile: Agree to use barrier contraception during treatment and for at least 3 months after the last dose of otuzumab or bendamustine or as required by guidelines established by the institution, whichever is longer. In addition, male patients must agree to have their partner use an alternative method of contraception (e.g., oral contraceptive, intrauterine device, barrier method, or spermicide)
14. For women who are not surgically sterilized: agree to use two appropriate methods of contraception, such as oral contraceptives, intrauterine devices, or barrier methods, with spermicide for at least 28 days before starting study drug, during treatment, and for at least 12 months after the last dose of otuzumab or bendamustine, or for the time required by the guidelines established by the study institution (whichever is longer)

Exclusion Criteria:

1. Mature B-cell lymphoma previously treated with chemotherapy, immunotherapy, or radiation therapy
2. Evidence of aggressive NHL transformation
3. Known hypersensitivity to any study drug
4. Known sensitive to murine products
5. Central nervous system or meningeal involvement by lymphoma
6. Contraindications to the investigational drug included in the study treatment regimen
7. Positive test results for chronic hepatitis B infection (defined as positive HBsAg serology)
8. Hepatitis C positive (hepatitis C virus [HCV] antibody serology)
9. HIV or Human T-Lymphocytic Leukemia Virus 1 (HTLV1) positive
10. Evidence of any serious, uncontrolled co-morbidities that could affect compliance with the study protocol or interpretation of results, including but not limited to significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmias, or unstable angina), or significant pulmonary disease (including history of obstructive pulmonary disease or bronchospasm);
11. Infection caused by known active bacteria, viruses, fungi, or other microorganisms (except fungal infection of the nail bed), or any major infection requiring intravenous antibiotics or hospitalization (completion of the entire course of antibiotics, except for neoplastic fever) within 4 weeks prior to enrollment
12. Previous history of malignancy other than lymphoma, unless the subject has a disease-free survival of ≥ 5 years
13. Pregnant or lactating women.
14. Participated in other clinical trials using drug interventions during the trial or within 28 days prior to Cycle 1 Corticosteroids within 4 weeks of enrollment, unless administered at a dose equivalent to ≤ 30 mg/day prednisone (within 4 weeks)

16. Past history of progressive multifocal leukoencephalopathy (PML) Vaccination with live vaccines within 28 days prior to start of treatment 18. History of solid organ transplantation 19. Presence of any serious disease or abnormality in the clinical laboratory test results that, in the opinion of the investigator, could make the patient unable to safely participate in and complete this study, or affect protocol compliance or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate(ORR) | 24 weeks
  Disease response evaluation after 6 cycles will be used to determine the overall remission rate

SECONDARY OUTCOMES:
Progression Free Survival | up to 4.5 years
  Progression free survival is defined as the time from the day in which the patient is enrolled to the date on which tumor progresses or the date on which the patient dies for any cause. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
Event-Free Survival | up to 4.5 years
  Event-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse, initiation of new anti-lymphoma therapy or death from any cause.
Complete Response Rate | 24 weeks
  Disease response evaluation after 6 cycles will be used to determine the overall remission rate
Overall survival | up to 4.5 years
  Overall survival will be measured from the date of inclusion to the date of death from any cause.
  Alive patients will be censored at their last date known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese
Locations (1):
- Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China